CLINICAL TRIAL: NCT07274072
Title: Hospital at Home Versus Inpatient Care: Costs and Effectiveness
Status: Recruiting | Type: Observational
Sponsor: Hospital at Home AG (Industry)
Collaborators: Klinik Hirslanden, Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-00482
Record Dates: First submitted 2025-09-22; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Costs and Cost Analysis; Effectiveness; Patient Satisfaction
Keywords: hospital at home; costs; clinical outcome; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital at Home Group: 100 participants treated in hospital at home
- Regular hospital group/"Brick and mortar group": 100 participants treated in the hospital

SUMMARY:
Background and Objectives Hospital at Home (HaH) delivers hospital-level treatment to acutely ill patients in their own homes, including daily medical and nursing visits, infusions, physiotherapy, and diagnostics. It bridges inpatient and outpatient care, working closely with hospitals, office-based physicians, home care services (Spitex), and therapy providers.

There are two main pathways:

Admission Avoidance: stable patients requiring hospitalization are admitted directly to HaH instead of an inpatient ward.

Early Supported Discharge: patients treated in hospital are discharged earlier than usual and transferred to HaH.

Evidence International studies show HaH to be safe and effective. Reviews report comparable mortality and rehospitalization, shorter hospital stays, and cost advantages. Admission avoidance is linked to trends toward lower mortality and costs. Research showed similar mortality but fewer rehospitalizations, longer treatment duration, and reduced risks of institutionalization, depression, and anxiety. HaH patients were older, with reduced daily living activities, yet care costs were on average USD 5,054 lower than inpatient care.

In Switzerland, the mean hospital stay in 2019 was 8 days (acute somatic: 5.2; psychiatry: 33.5).

Study Hypotheses

HaH can be delivered at equal or lower cost than regular hospitalization.

HaH care is safe, with few complications, and yields high patient satisfaction.

Study Objective To demonstrate that hospital-equivalent home treatment of acutely ill patients is effective, appropriate, cost-efficient (according to Swiss WZW criteria), safe, and associated with high satisfaction and low complication rates compared with inpatient care.

Endpoints

Primary: Costs - HaH vs. inpatient care at Hirslanden Clinic, using REKOLE® cost accounting.

Secondary: Mortality, therapy type, monitoring, diagnostics, rehospitalization, complications, satisfaction, patient-reported outcomes, length of stay, referrals to nursing homes, follow-up after discharge, ED visits, rehabilitation referrals, and home care type.

DETAILED DESCRIPTION:
1. BACKGROUND AND SIGNIFICANCE OF THE STUDY

   The Hospital at Home concept enables hospital-equivalent treatment of acutely ill patients requiring hospitalization in their own homes. Treatment is carried out as in a regular hospital, with daily visits by physicians and nurses. In addition to disease management, including infusion therapies, home-based physiotherapy and diagnostic procedures such as blood and urine testing, ultrasound, and electrocardiography are provided.

   This positions Hospital at Home at the interface between traditional inpatient and outpatient care, complementing the existing services of hospitals, office-based physicians, home care organizations (Spitex), physiotherapy, and occupational therapy through a structured treatment process at the patient's home. Care is not provided in isolation but in cooperation with the aforementioned established institutions.

   Two referral pathways into Hospital at Home can be distinguished:

   Admission Avoidance: eligible patients in stable general condition with an acute illness that would normally require hospitalization are admitted directly into Hospital at Home instead of inpatient care and treated equivalently at home.

   Early Supported Discharge: patients already treated in a regular hospital and in good general condition are discharged earlier than usual and transferred to Hospital at Home, where treatment is completed.

   Hospital at Home has been investigated in various international studies. A review found, patients assigned to Hospital at Home via early supported discharge showed comparable mortality and rehospitalization rates and shorter hospital stays. Patients admitted via admission avoidance showed a trend towards lower mortality and costs and comparable rehospitalization rates.

   Further research found similar mortality rates between Hospital at Home and regular inpatients, but lower rehospitalization rates and longer treatment durations in the Hospital at Home group. It also showed lower risk of institutionalization in long-term care facilities, as well as a reduced risk of depression and anxiety.

   A retrospective observational study from New York, USA, showed, that Hospital at Home patients were on average older and showed reduced activities of daily living. The costs of Hospital at Home care were on average USD 5054 lower than those of comparable inpatients.

   In Switzerland in 2019, the average length of stay across all hospital sectors was 8.0 days, with the shortest in acute somatic care (5.2 days) and the longest in psychiatry (33.5 days).
2. PROJECT OBJECTIVES AND DESIGN 2.1 Hypotheses and Primary Study Objective

Hypothesis 1 Care through Hospital at Home can be delivered at equivalent or lower cost compared to regular hospitalization.

Hypothesis 2 Hospital at Home care is safe for patients, associated with few complications, and yields high patient satisfaction.

Study Objective Our study aims to demonstrate that hospital-equivalent treatment of acutely ill patients at home is effective, appropriate, and cost-efficient (according to the Swiss WZW criteria) and, compared with regular inpatient care, is safe, associated with low complication rates, and achieves high patient satisfaction.

2.2 Primary and Secondary Endpoints

Primary Endpoint:

Costs: Treatment in Hospital at Home can be cost-equivalent or more cost-effective compared to regular inpatient care. Patient data from Hospital at Home AG will be compared with patient data from regular inpatients at Hirslanden Clinic. Costs, or billable tariffs, will be considered based on cost accounting according to REKOLE®.

Secondary Endpoints (as defined in section 3.3 "Additional Study Variables"):

Mortality

Type of therapy

Type of monitoring

Type and frequency of diagnostics

Rehospitalization during and after treatment

Complications and complication rates

Patient satisfaction

Patient-related outcomes

Length of stay

Referrals to nursing homes or long-term care after discharge

Follow-up with general practitioner or specialist after discharge

Emergency department visits during treatment and after discharge

Referral to rehabilitation clinics after discharge

Type of home care after discharge

ELIGIBILITY:
Inclusion Criteria:

* Inpatients in the hospital or patients in Hospital at Home care
* Age ≥ 18 years
* Admission due to a typical Hospital at Home diagnosis (mild to moderate inflammatory and infectious diseases of the lungs, urinary tract, gastrointestinal tract, heart, and skin; exacerbated chronic obstructive pulmonary disease; exacerbation of chronic heart failure; wounds; bleeding/anemia; dehydration; deterioration of general condition in multimorbid patients; infection-related complications in oncological patients; psychiatric problems including delirium; metabolic or autoimmune diseases; orthopedic patients; pain exacerbations of any cause; palliative patients up to and including terminal situations)
* Patients without severe cognitive impairment or dysfunction who are capable of providing informed consent and/or completing the questionnaire
* Patients with sufficient proficiency in written and spoken German and/or English

Exclusion Criteria:

* Inpatient admission for other reasons
* Refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 participants total, 100 from the regular hospital ("brick and mortar"), 100 from Hospital at Home. Patients from 18years of age upwards with a disease treated in the hospital or in hospital at home.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Costs | 1 year or until the total of 200 participants are included
  Comparison of cost of treatment in Hospital at Home vs. regular hospital ("brick and mortar"). Data will be collected via financal data of both groups, 100 patients from the regular hospital (Klinik Hirslanden Zurich) and 100 patients from Hospital at Home AG (Zollikon)

SECONDARY OUTCOMES:
Effectiveness (clinical outcome) | 1 year or until the total of 200 participants are included
  Measure of how effective the treatment in Hospital at Home vs. regular hospital ("brick and mortar") is. The clinical outcome will be measured by: Mortality up to 30 days after discharge, emergency-admission up to 30 days after discharge, readmission to the hospital/H@H up to 30 days after discharge, GP-consultation up to 30 days after discharge, specialist-consultation up to 30 days after discharge, admission to nursing home up to 30 days after discharge. Data will be collected through patient data, collected via clinical information system and phone calls to the patient 30 days after discharge.
Effectivness (complications) | 1 year or until the total of 200 participants are included
  Measure of how effective the treatment in Hospital at Home vs. regular hospital ("brick and mortar") is. The clinical outcome will be measured by measuring the number and kind of complication. We will collect data regarding number of falls, (up to 30 days after discharge), number of new infections during treatment, development of bedsores during treatment (yes/no), development of delirium during treatment (yes/no), thrombosis during treatment (yes/no). Data will be collected through patient data, collected via clinical information system and phone calls to the patient 30 days after discharge.
Patient satisfaction | 1 year or until the total of 200 participants are included
  How satisfied are the patients treated in Hospital at Home compared to patients treated in the regular hospital ("brick and mortar"), measured by patient questionnaires. First questionnaire (patient satisfaction) consists of 8 questions each reaching from 0-5 points (0 = worst, 5 = best) regarding overall assessment, recommendation of service, assessment by relatives, competencies of nurses, competencies of doctors, quality of hotline, satisfaction with communication/flow of information and safety. Second questionnaire ist the PROMIS Globla health 10 consisting of 10 questions, first 9 reaching from 1-5, last question reaching from 0-10 points. The questions assess global well-being, quality of life, physical and psychological well-being, satisfaction with level of activity, handling of everyday activities, handling of everyday phsysical tasks, mental problems, tiredness, pain. Data will be collected through patient data, collected via clinical information system and phone calls.

OTHER OUTCOMES:
patient data | 1 year or until the total of 200 participants are included
  Data regarding demographics including name, date of birth, age, sex, language, distance hospital to home, date of death, date of admission/discharge, length of stay, ICD-codes, -chapters, major diagnostic chapters, type of insurance, billing, referrer, living situation (alone yes/no), care situation (independent, nursing home), nr of drugs ad admission/30d post discharge, polypharmacy (defined as >5 drugs at admission), nr of chronic comorbidities, Charlson comorbidity score/-10 year survival rate, cognitive impairment (yes/no), i.v.-medication during treatment (yes/no, duration), monitoring (yes/no, duration), nr of hotline calls/ringing of nurse, nr of doctor/nurses visits, nr of ecg/sonography/xray/expert consultation, yes/no of physiotherapy/O2-substitution.
  Data will be collected through patient data, collected via clinical information system and phone calls to the patient 30 days after discharge.
result of first blood sample | 1 year or until the total of 200 participants are included
  Collection of results of first blood sample, taken at admission to hospital/H@H. Collection of white blood cell count G/l, hemoglobin g/l, CRP mg/l, natrium mmol/l, potassium mmol/l, creatinine umol/l, GFR ml/min/1.73m2, ALT U/l. Data will be collected through patient data, collected via clinical information system and phone calls to the patient 30 days after discharge.
first vital signs measured at admission | 1 year or until the total of 200 participants are included
  Collection of values of first vital sign measurement at admission. Collection of SpO2 in %, body temperature in °C, blood pressure in mmHg, respiratory rate in x/min. Data will be collected through patient data, collected via clinical information system and phone calls to the patient 30 days after discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital at Home AG, Zollikon, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Would be interesting to compare data with other Hospital at Home programs, but no plans are yet made.

REFERENCES:
- [Result] Leong MQ, Lim CW, Lai YF. Comparison of Hospital-at-Home models: a systematic review of reviews. BMJ Open. 2021 Jan 29;11(1):e043285. doi: 10.1136/bmjopen-2020-043285. PMID 33514582